CLINICAL TRIAL: NCT03231631
Title: Efficacy Of An Education Plan And Adherence Follow-Up To The Exercise In Patients With Angioplasty And Implantation Of Coronary Stent, Measured With Hdl And Met In A Cardiac Rehabilitation Unit - Random Triple Blind Clinical Trial
Brief Title: Efficacy Of An Education Plan And Adherence Follow-Up To The Exercise In Patients With Angioplasty And Stent Coronary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica de Occidente S.A (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2017-07-01; First posted 2017-07-27 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Patient Adherence
Keywords: Exercise; Education; Stents; Angioplasty; Cardiac Rehabilitation; Cholesterol, HDL; Metabolic Equivalent
MeSH Terms: conditions — Patient Compliance; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education plan and adherence to exercise (Experimental): * Educational talk about the importance of nutrition and exercise as an important strategy to change cardiovascular risk factors at the start of the study.
  * It will be sent via text, whatsapp, and / or e-mail on a weekly basis three text messages that remind them of the importance of doing the exercise and how often they should do it, it will be a predetermined text.
  Interventions: Behavioral: Education plan and adherence to exercise
- Control (No Intervention): The blood sample will be taken for the collection of serum HDL and the aerobic capacity test measured in MET will be recorded at the beginning of the study.
  A survey will be conducted at week 12 of monitoring where adherence to exercise is measured during the 12-week study.

INTERVENTIONS:
Behavioral: Education plan and adherence to exercise — * Send text messages with motivational sense at any time of the day, every 3 or 4 days.
  * They will be given the option of performing directed exercise at the cardiac rehabilitation center.
  * It will be recorded in an Excel table every time that text is sent to the patient.
  * At the beginning and monthly, a brochure will be sent out explaining how physical activity is performed at home in case you can not walk.
  * A monthly survey will be applied where the adherence to the exercise during the previous month is measured.
  * These activities will be carried out for 12 weeks. At the end of week 12, patients will be referred to the cardiac rehabilitation unit in order to perform the aerobic capacity test again.
  Arms: Education plan and adherence to exercise

SUMMARY:
Cardiovascular diseases are a leading cause of death worldwide. Some of the risk factors that have been identified are considered as be non-modifiable and modifiable. Among the non-modifiable, gender, age, race, family history and pathological antecedents such as diabetes and hypertension among others are taken into account. The modifiable factors are weight, abdominal circumference, habits such as smoking, alcohol consumption, diet and especially the EXERCISE.

In order to modify these risk factors, patients are submitted to a strategy of health promotion, disease prevention, pharmacological treatments, non-invasive and invasive treatments such as cardiac catheterization, balloon coronary angioplasty and / or stent implantation, cardiovascular surgeries etc. However, one of the most important strategies that should be of great importance is to involve the patient and his family in these treatments through education and follow-up strategies whether it is through the telephone, home visit, e-mail, messages, etc. In this way, the patient is brought to a state of self-determination and self-awareness that leads him to perform physical activity routinely so he can change his cardiovascular risk factors and become a patient adherent to exercise or any other treatment. This is where the importance of exercise or aerobic physical activity is emphasized, as it is a low-cost activity that can be performed by any type of patient, and that results are easily observed in physical and physiological changes that can be objectively measurable, such as the levels in serum lipid profile (cholesterol, triglycerides, LDL and HDL), or cardiovascular function tests such as stress tests with METs indicating increased aerobic capacity (Improvement in ability to withstand a stress test).

Therefore, the purpose of this study is to submit a group of patients to an education and telephone follow-up plan, emphasizing on the importance of performing physical activity with the appropriate intensity and frequency so that they can include it within their daily routine by itself and ensure "the adherence to physical activity".

Physiological changes that these patients may present as a consequence of the acquired routine physical activity by being subject to the education and telephone follow-up plan of this research will be measured with serum HDL levels in a clinical laboratory test and MET in a stress test.

DETAILED DESCRIPTION:
According to the population of the cardiac rehabilitation center of the Private IPS of Cali, it will be analyzed by the program coordinator (Cardiac Rehabilitation Center) who are the patients that finished the 36 sessions or finished their rehabilitation treatment scheme and that will become potential candidates for the study.

If the patient is considered a candidate to enter the study, an interview will be made to explain what the study is about and to verify whether or not he wishes to participate, without indicating to which group he will belong (follow-up or control). If the patient agrees to participate in the study, the process of signing the informed consent and the application of the clinical trail where the basic patient information necessary for the study entrance is collected.

Once the informed consent is signed, the patient is given a physical examination of his clinical and physical condition (anthropometric parameters - exercise test) at the beginning of the exercise, which consists of physical ergonomic tests (exercise test).

The test was performed from a symptom-limited ergometry in a treadmill stress test kit. The Bruce protocol was used in the treadmill, which started after a warm-up period of three minutes. During the test, continuous electrocardiographic monitoring and blood pressure measurements were performed with a blood pressure monitor and heart rate monitor. The test was terminated by the onset of fatigue, severe dyspnea, dizziness or when the patient reached the highest heart rate expected for age, accompanied by the medical internist of the private IPS program.

Additionally, a medical order is given with the respective recommendations (identifying that the patient belongs to the study), for the collection of HDL blood in the clinical laboratory hired for this purpose, in this way, the clinical laboratory does not perform authorization requirements or that the patient has obstacles with HDL taking).

Allocation concealment: Once the physical tests and anthropometric parameters were completed and the clinical survey was applied, the information was stored in a closed envelope and a consecutive number was assigned according to the order of the exercise. The envelopes were sent to the person responsible for the implementation of the tracking plan that according to the order and the consecutive number will be added on the database.

The randomization of the groups is done in a pre-established template as follows: Simple random sampling with Excel, a list is processed in the table of the study database and where variables are collected, the numbering of anger from 1 to 80 according to the number of patients required to enter the study, apply a simple randomization formula and a different Excel spreadsheet, up to number 40 (the amount corresponding to the entire follow-up group (group A) and control group B)), the numbers that have resulted from this randomization are those assigned to the follow-up group.

In this way, when patients are registered in the database in the numerical order in the envelope, it is automatically assigned according to the randomization of the group to which the patient belongs (Follow-up or control).

After the patients are entered into the database of data collection and variables, the patients belonging to the follow-up group (already marked according to previous randomization) are separated and sent to the responsible nursing assistant with the purpose of starting the established monitoring plan, such the activity must be registered in an Excel table where the control and registration of the same will be carried out.

Once the nursing assistant responsible for the implementation of the follow-up plan will proceed to carry out her activities as follows.

She will check the number of patients entering the study, check the date of entry and date of completion, confirm that all patients have cellphone and land numbers where they can be located, in addition to their residence address and email.

She will verify that the follow-up boxes for each patient are completed, which are performed twice weekly for a total of 24 follow-ups or 12 weeks, duration of the follow-up plan.

She will start with phone calls, text messages and email according to the established schedule in the work template or tracking log format.

In each follow-up box for each patient it will record the type of activity that performed, call, text message or email where she sent the necessary recommendations for patients to exercise.

Once the follow-up and the time are completed, the list of the patients who have completed the data collection will be sent to the program to schedule the second studies in HDL and Exercise TEST in The Center for Cardiac Rehabilitation.

An exercise adherence survey will be applied once the patient goes on week 6 or follow-up number 12 in order to measure adherence to exercise by the patient. This result will be processed in the tracking table, the applied surveys will be saved in a file other than Excel.

Once the follow-up is completed, the patient will stop calling and the record will be handed over to the person responsible for collecting data.

In the control group, according to the dates of entry to the study in week 6 related to the order of admission, a survey of adherence to the exercise will be applied by an administrative assistant who will keep a record of the same in a separate file and the respective result.

As the 12-week study period ends, the cardiac rehabilitation nurse assistant will receive the names of the patients and their respective phones from both the follow-up group and the control group without having any group marking to which one they belong, so that the second physical test or exercise test is performed and their respective order of clinical laboratory HDL is given.

Through email, the laboratory will be requested to deliver physically and in a sealed envelope all the results of tests performed to the patients that belong to the study. These results will be delivered to the database manager and registry of variables.

All the documentation that as a result of the study, will be guarded by the person in charge of the management of the database and registration of variables.

The person in charge of the database and registry of variables is the one who will inform the moment in which the study has finished. Subsequently, the information will be organized and the data will be given to the methodological adviser in order to organize, process and analyze the statistical information as a result of it.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative subjects of angioplasty with implantation of coronary stent
* Age between 35 and 65
* Subjects with ability to perform the aerobic capacity test
* Subjects culminating the cardiac rehabilitation program (3 months)

Exclusion Criteria:

* Active phase of any acute disease
* Poor adherence to the rehabilitation program (failure to comply with appointments or with the recommendations given)
* Patient with cardiovascular decompensation (unstable angina)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Adherence to exercise | Measured at the end of the 12 week monitoring
  Perform routine physical activity as a principle of self-determination and convert it into a healthy lifestyle or habit

SECONDARY OUTCOMES:
Change in HDL levels and MET | Measured at baseline HDL and MET and at the end of the 12 week monitoring
  Change in HDL level and MET as the difference between baseline HDL and MET and final HDL and MET

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ávila, PT, Principal Investigator — Clínica de Occidente S.A
Locations (1):
- Juan Carlos Avila, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eden KB, Orleans CT, Mulrow CD, Pender NJ, Teutsch SM. Does counseling by clinicians improve physical activity? A summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2002 Aug 6;137(3):208-15. doi: 10.7326/0003-4819-137-3-200208060-00015. PMID 12160371
- [Background] Ilarraza-Lomeli H. [Cardiopulmonary exercise testing]. Arch Cardiol Mex. 2012 Apr-Jun;82(2):160-9. Spanish. PMID 22735657
- [Background] Ilarraza Lomeli H, Herrera Franco R, Lomeli Rivas A, Zavala Ramirez J, Martinez Ramirez L, Ramos Becerril FJ, Romo Escamilla RE, Pacheco Beltran N, Alonso Sanchez J, Mendoza Diaz PM, Alvarez Cerro M, Cassaigne Guasco ME, Mayela Munoz Gutierrez LM. [National Registry of Cardiac Rehabilitation Programs in Mexico]. Arch Cardiol Mex. 2009 Jan-Mar;79(1):63-72. Spanish. PMID 19545077
- [Background] Antunez de la Rosa Mdel R, Jimenez y Villegas Mdel C. [Nurses' participation in heart rehabilitation]. Arch Cardiol Mex. 2002 Jan-Mar;72 Suppl 1:S247-53. Spanish. PMID 12001856
- [Background] Gomez LF, Duperly J, Lucumi DI, Gamez R, Venegas AS. [Physical activity levels in adults living in Bogota (Colombia): prevalence and associated factors]. Gac Sanit. 2005 May-Jun;19(3):206-13. doi: 10.1157/13075953. Spanish. PMID 15960953
- [Background] Pollock JL. Low HDL cholesterol levels. N Engl J Med. 2006 Jan 26;354(4):417-9; author reply 417-9. No abstract available. PMID 16444813
- [Background] Médicas FDEC, Del R, Hdl C, Carol A, Rojas J. Departamento de Postgrado ANTE EL EJERCICIO FISICO AEROBICO Y ANAEROBICO ".
- [Background] Hernán, V., William, R., Jaime, B., & Jorge R. Fundamentos de medicina. Cardiología. Sexta edic. Biológicas C para I, editor. 2002.
- [Background] Claudia V. Anchique M, ; Carmen Pérez-Terzic MD., PhD.; Francisco López-Jiménez, MD., MSc. ; Mery Cortés-Bergoderi M. Estado actual de la rehabilitacion cardiovascular en Colombia. 2010;18(6):305-15. Available from: http://www.discapacidadcolombia.com/Estadisticas.htm
- [Background] Global status report on noncommunicable diseases. Who. 2010;ISBN: 978 92 4 156422 9.
- [Background] Velasquez G. [Global access to medications in the actual international context ]. Biomedica. 2011 Jun;31(2):162-3. doi: 10.1590/S0120-41572011000200001. No abstract available. Spanish. PMID 22159530
- [Background] Porqueres IM. Rol del fisioterapeuta en el marco de la rehabilitación cardíaca. Fisioterapia [Internet]. 2003;25(3):170-80. Available from: http://db.doyma.es/cgi-bin/wdbcgi.exe/doyma/mrevista.fulltext?pident=13049838\nhttp://www.sciencedirect.com/science/article/pii/S0211563803730533
- [Background] Leon AS, Franklin BA, Costa F, Balady GJ, Berra KA, Stewart KJ, Thompson PD, Williams MA, Lauer MS; American Heart Association; Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention); Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity); American association of Cardiovascular and Pulmonary Rehabilitation. Cardiac rehabilitation and secondary prevention of coronary heart disease: an American Heart Association scientific statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity), in collaboration with the American association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2005 Jan 25;111(3):369-76. doi: 10.1161/01.CIR.0000151788.08740.5C. PMID 15668354
- [Background] Velasco JA, Cosin J, Maroto JM, Muniz J, Casasnovas JA, Plaza I, Abadal LT. [Guidelines of the Spanish Society of Cardiology for cardiovascular disease prevention and cardiac rehabilitation]. Rev Esp Cardiol. 2000 Aug;53(8):1095-120. Spanish. PMID 10956605
- [Background] Clinicoquir HD, Deportiva M. Influencia del ejercicio físico sobre algunos factores de riesgo de la cardiopatía isquémica. 1998;17(3):214-21.
- [Background] Caramés AZI. Impacto de un programa de rehabilitación cardiovascular en perfil antropométrico, alimentario y lipídico en pacientes con enfermedad coronaria. 2012;
- [Background] Pico cjr. respuesta del colesterol hdl ante el ejercicio físico aeróbico y anaeróbico".
- [Background] Tseng ML, Ho CC, Chen SC, Huang YC, Lai CH, Liaw YP. A simple method for increasing levels of high-density lipoprotein cholesterol: a pilot study of combination aerobic- and resistance-exercise training. Int J Sport Nutr Exerc Metab. 2013 Jun;23(3):271-81. doi: 10.1123/ijsnem.23.3.271. Epub 2012 Nov 19. PMID 23166203
- [Background] Manuel Wong, Miriam García, Adriana García SC. Resultados del Programa de Rehabilitación Cardíaca Fase II , desarrollado por el Centro Nacional de Rehabilitación , Costa Rica. 2011;
- [Background] Janssen V, De Gucht V, van Exel H, Maes S. A self-regulation lifestyle program for post-cardiac rehabilitation patients has long-term effects on exercise adherence. J Behav Med. 2014 Apr;37(2):308-21. doi: 10.1007/s10865-012-9489-y. Epub 2013 Jan 19. PMID 23334387
- [Background] SÍNDROME CORONARIO AGUDO CON ELEVACIÓN DEL ST. Rev Colomb Cardiol. 2007;17(03):186-317.
- [Background] Pavy B, Iliou MC, Verges-Patois B, Brion R, Monpere C, Carre F, Aeberhard P, Argouach C, Borgne A, Consoli S, Corone S, Fischbach M, Fourcade L, Lecerf JM, Mounier-Vehier C, Paillard F, Pierre B, Swynghedauw B, Theodose Y, Thomas D, Claudot F, Cohen-Solal A, Douard H, Marcadet D; Exercise, Rehabilitation Sport Group (GERS); French Society of Cardiology. French Society of Cardiology guidelines for cardiac rehabilitation in adults. Arch Cardiovasc Dis. 2012 May;105(5):309-28. doi: 10.1016/j.acvd.2012.01.010. Epub 2012 Apr 16. No abstract available. PMID 22709472
- [Background] Piepoli MF, Corra U, Benzer W, Bjarnason-Wehrens B, Dendale P, Gaita D, McGee H, Mendes M, Niebauer J, Zwisler AD, Schmid JP; Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Secondary prevention through cardiac rehabilitation: from knowledge to implementation. A position paper from the Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Eur J Cardiovasc Prev Rehabil. 2010 Feb;17(1):1-17. doi: 10.1097/HJR.0b013e3283313592. PMID 19952757
- [Background] European Association of Cardiovascular Prevention and Rehabilitation Committee for Science Guidelines; EACPR; Corra U, Piepoli MF, Carre F, Heuschmann P, Hoffmann U, Verschuren M, Halcox J; Document Reviewers; Giannuzzi P, Saner H, Wood D, Piepoli MF, Corra U, Benzer W, Bjarnason-Wehrens B, Dendale P, Gaita D, McGee H, Mendes M, Niebauer J, Zwisler AD, Schmid JP. Secondary prevention through cardiac rehabilitation: physical activity counselling and exercise training: key components of the position paper from the Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Eur Heart J. 2010 Aug;31(16):1967-74. doi: 10.1093/eurheartj/ehq236. Epub 2010 Jul 19. PMID 20643803
- [Background] Pulmonary rehabilitation: joint ACCP/AACVPR evidence-based guidelines. ACCP/AACVPR Pulmonary Rehabilitation Guidelines Panel. American College of Chest Physicians. American Association of Cardiovascular and Pulmonary Rehabilitation. Chest. 1997 Nov 5;112(5):1363-96. No abstract available. PMID 9367481
- [Background] Wenger NK. Current status of cardiac rehabilitation. J Am Coll Cardiol. 2008 Apr 29;51(17):1619-31. doi: 10.1016/j.jacc.2008.01.030. PMID 18436113
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Aznar S, Webster T. Actividad física y salud en la infancia y la adolescencia: Guía para todas las personas [Internet]. 2006. Available from: http://www.msssi.gob.es/ciudadanos/proteccionSalud/adultos/actiFisica/docs/ActividadFisicaSaludEspanol.pdf
- [Background] Hillsdon M, Foster C, Thorogood M. Interventions for promoting physical activity. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003180. doi: 10.1002/14651858.CD003180.pub2. PMID 15674903
- [Background] Richards J, Hillsdon M, Thorogood M, Foster C. Face-to-face interventions for promoting physical activity. Cochrane Database Syst Rev. 2013 Sep 30;2013(9):CD010392. doi: 10.1002/14651858.CD010392.pub2. PMID 24085592